CLINICAL TRIAL: NCT06141304
Title: A Single Arm Study of Using Plerixafor Plus Donor Lymphocyte Infusion in the Treatment of Patients With Relapsed Acute Leukemia After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Plerixafor Plus Donor Lymphocyte Infusion for Relapsed Acute Leukemia After Allo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, SuJun Gao, Professor, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLEU
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Relapsed Adult ALL; Relapsed Adult AML
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — plerixafor

STUDY DESIGN:
Intervention Model Description: Plerixafor plus donor lymphocyte infusion for patients with relapsed acute leukemia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plerixafor plus DLI (Experimental): DLI will be given to the participants three days after chemotherapy, and plerixafor will be administrated ten days post DLI.
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Plerixafor was injected subcutaneously to participants twice per day for five consecutive days ten days post DLI.
  Other Names: AMD3100

SUMMARY:
Acute leukemia, including acute myeloid leukemia (AML) and acute lymphoblastic leukemia (ALL), is the subtype of leukemia with the highest mortality, and leukemia relapse caused by the protective bone marrow microenvironment is the main cause of treatment failure. The chemokine receptor CXCR4 plays a crucial role in the homing and settling of leukemia cells into the bone marrow. Preclinical study of the investigators demonstrates that CXCR4 blockade can mobilize leukemia cells from their protective bone marrow microenvironment to periphery, thereby significantly enhancing the killing effect of allogeneic lymphocytes against leukemia cells. This study aims to preliminarily evaluate the efficacy and safety of donor lymphocyte infusion (DLI) plus CXCR4 antagonist plerixafor in the treatment of relapsed acute leukemia patients after allogeneic hematopoietic stem cell transplantation (allo-HSCT) through a prospective single arm study. The results may preliminarily confirm the effectiveness and safety of DLI combined with plerixafor in the treatment of recurrent acute leukemia patients after allo-HSCT, providing a reference basis for further research.

DETAILED DESCRIPTION:
Patients with relapsed acute leukemia post allo-HSCT will be screened for the eligibility of this clinical trial. The participants will receive chemotherapy to reduce leukemia burden followed by DLI three days later. Ten days post DLI, plerixafor will be administrated to the participants (subcutaneous injection, twice per day) for a consecutive five days. The second round of DLI plus plerixafor will be given if the participants achieving partial remission or complete remission with positive minimal measurable disease. Short-term responses and long-term outcomes will be evaluated and safety of this therapeutic regimen will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patients is ≥ 14 and ≤ 60 years old;
* Those with relapsed acute leukemia after allo-HSCT with bone marrow blasts less than 50%;
* The expected survival exceeds 3 months;
* At least 100 days post transplantation, and the immunosuppressants were discontinued;
* Those with no significant abnormalities of the main organ function: creatinine ≤ 176.8 μ Mol/L, bilirubin ≤ 51.3 μ Mol/L, aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the normal upper limit;
* Sign an informed consent form.

Exclusion Criteria:

* Those with patient-specific human leukocyte antigen (HLA) loss at relapse;
* Those with active graft-versus-host disease;
* Those with severe infection;
* Those with organ function failure;
* Those with an Eastern Cooperative Oncology Group (ECOG) score more than 2 points;
* Those who are allergic to experimental drugs;
* Those who use other anti-leukemia therapies, such as radiotherapy, cellular immunotherapy, or Chinese medical herbs;
* Those participate in other clinical trials simultaneously;
* Those having mental illness or other illnesses that cannot fully comply with treatment or follow-up requirements;
* Those with extramedullary leukemia;
* Those with other conditions that researchers evaluate who are not proper to participate in this clinical trial.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Remission rates of the enrolled participants | Three months
  The remission rates of the participants include complete remission rate, partial remission rate, and overall response rate.

SECONDARY OUTCOMES:
Disease-free survival (DFS) of the enrolled participants | Twelve months
  DFS is defined from achievement of complete remission to disease relapse.
Overall survival of the enrolled participants | Twelve months
  DFS is defined from enrollment to death, last contact, or end of this clinical trial.
Number of participants with acute and chronic graft-versus-host disease (GVHD) | Twelve months
  Any grade of acute and chronic GVHD of the participants will be recorded. The acute GVHD will be assessed by MAGIC guidelines and chronic GVHD will be assessed by National Comprehensive Cancer Network (NCCN) guidelines.
Number of participants with non-relapse mortality | Twelve months
  Non-relapse mortality (NRM) is defined as any cause of death without leukemia relapse.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | One month after treatment
  Treatment-related adverse events will be assessed by CTCAE v5.0, including hematological and non-hematological adverse events. However, the occurrence of GVHD is not included.

CONTACTS AND LOCATIONS:
Overall Officials: Long Su, PhD, Study Director — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China